CLINICAL TRIAL: NCT04145557
Title: The Effect of Periodontal Treatment With 980nm Diode Laser on the State of Periodontium and Inflammatory Markers in Generally Healthy Patients and Patients After Myocardial Infarction
Brief Title: 980nm Diode Laser in the Treatment of Periodontal Disease in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Renata Samulak, Principal investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB-0012/06/12 KB-0012/09/1
Record Dates: First submitted 2019-10-24; First posted 2019-10-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction; Periodontal Diseases
Keywords: periodontitis; diode laser; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Periodontal Diseases; Periodontitis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skaling root planing (Placebo Comparator)
  Interventions: Device: scaling root planing
- skaling root planing and diode laser (Active Comparator)
  Interventions: Device: diode laser 980nm

INTERVENTIONS:
Device: diode laser 980nm — Procedure: Periodontal therapy with laser Scaling, root planning, oral hygiene instruction and diode laser 980nm treatment of periodontal pockets
  Arms: skaling root planing and diode laser
Device: scaling root planing — scaling and root planing
  Arms: skaling root planing

SUMMARY:
The study will cover 80 patients under 70 years of age. Initially they will be assigned to three groups: patients generally healthy with periodontitis (P), patients after myocardial infarction with periodontitis (CP) and patients generally healthy with a healthy periodontium (H). Periodontal examination will be performed before treatment, 2 weeks and 3 months after the treatment with a Williams probe calibrated at intervals 1-2-3-5-7-8-9-10mm. Pocket depth (PD), clinical loss of the attachment (CAL) bleeding on probing (BOP), plaque control record (PCR) measurements will be performed. Clinical data will be collected at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) of the designated study teeth. PD will be measured in millimeters from the free gingival margin to the base of the probable pocket using a periodontal probe. The presence of BOP will be determined as being present or absent (+/-) within 30 seconds after probing. CAL will be defined as the distance from the cementoenamel junction to t the base of the probable pocket .

Patients within CP and P groups will be randomly assigned to one of the two groups (study group and control group) and an later visit will be scheduled.

Before treatment, teeth will be rinsed and the study areas will be isolated with cotton rolls and dried gently. Supragingival plaque will then be removed with a sterile curret without coming into contact with the gingiva. GCF samples will be collected from the deepest single root tooth pockets previously identified. The sample will be collected from the deepest pocket using the Periopaper strips (OraflowInc., USA). Before collecting the material, the teeth will be insulated with cotton swabs. The teeth will then be dried with air. The strips will be placed in pockets until a slight resistance is perceived, and they will be left in place for 30 seconds and then transferred to Periotron 8000 (OraflowInc., USA) for the determination of fluid volume. Strips contaminated by bleeding will be discarded.

Next, each strip will be inserted into the Eppendorff tube and sent to the laboratory at the Medical Analytics Department of PUM in Szczecin for further analysis. The volume of the gingival fluid will be given in μl, in accordance with the conversion of values displayed as a reading on the device.

The microbiological examination (via Real-PCR method) for the presence of pathogenic bacteria for periodontium will be performed using commercial standard sets PET-MIP deluxe ® (MIP Pharma). Samples will be taken from the patient's deepest periodontal pocket. After isolation of the examined tooth from the access of saliva, sterile paper will be placed inside the pocket for 10 seconds following transfer to the transport containers included in the PET-Mip deluxe ® kits and sent to the MIP-Pharma laboratory in St. Ingbert in Germany.

In the control and study group, supra and subgingival scaling and root smoothing with Gracey currets will be performed. Individual oral hygiene instructions will also be given to each patient. In addition laser therapy of the pockets with a 980nm diode laser will be carried out in the study group.

The levels of TC, LDL, HDL, TG, hsCRP, leukocytes, fibrinogen, OB, IL-6, AST, ALT in the peripheral blood will be marked three times (before treatment, 2 weeks and 3 months post treatment). For this purpose, the blood will be taken from the superficial veins of the forearm and sent for further analysis at the Medical Analytics Department of PUM in Szczecin.

DETAILED DESCRIPTION:
The study will cover 80patients under 70 years of age. Initially they will be assigned to three groups: patients generally healthy with periodontitis (P), patients after myocardial infarction with periodontitis (CP) and patients generally healthy with a healthy periodontium (H). Periodontal examination will be performed before treatment, 2 weeks and 3 months after the treatment with a Williams probe calibrated at intervals 1-2-3-5-7-8-9-10mm. Pocket depth (PD), clinical loss of the attachment (CAL) bleeding on probing (BOP), plaque control record (PCR) measurements will be performed. Clinical data will be collected at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) of the designated study teeth. PD will be measured in millimeters from the free gingival margin to the base of the probable pocket using a periodontal probe. The presence of BOP will be determined as being present or absent (+/-) within 30 seconds after probing. CAL will be defined as the distance from the cementoenamel junction to t the base of the probable pocket .

Patients within CP and P groups will be randomly assigned to one of the two groups (study group and control group) and an later visit will be scheduled.

Before treatment, teeth will be rinsed and the study areas will be isolated with cotton rolls and dried gently. Supragingival plaque will then be removed with a sterile curret without coming into contact with the gingiva. GCF samples will be collected from the deepest single root tooth pockets previously identified. The sample will be collected from the deepest pocket using the Periopaper strips (OraflowInc., USA). Before collecting the material, the teeth will be insulated with cotton swabs. The teeth will then be dried with air. The strips will be placed in pockets until a slight resistance is perceived, and they will be left in place for 30 seconds and then transferred to Periotron 8000 (OraflowInc., USA) for the determination of fluid volume. Strips contaminated by bleeding will be discarded.

Next, each strip will be inserted into the Eppendorff tube and sent to the laboratory at the Medical Analytics Department of PUM in Szczecin for further analysis. The volume of the gingival fluid will be given in μl, in accordance with the conversion of values displayed as a reading on the device.

The microbiological examination (via Real-PCR method) for the presence of pathogenic bacteria for periodontium will be performed using commercial standard sets PET-MIP deluxe ® (MIP Pharma). Samples will be taken from the patient's deepest periodontal pocket. After isolation of the examined tooth from the access of saliva, sterile paper will be placed inside the pocket for 10 seconds following transfer to the transport containers included in the PET-Mip deluxe ® kits and sent to the MIP-Pharma laboratory in St. Ingbert in Germany.

In the control and study group, supra and subgingival scaling and root smoothing with Gracey currets will be performed. Individual oral hygiene instructions will also be given to each patient. In addition laser therapy of the pockets with a 980nm diode laser will be carried out in the study group.

The levels of TC, LDL, HDL, TG, hsCRP, leukocytes, fibrinogen, OB, IL-6, AST, ALT in the peripheral blood will be marked three times (before treatment, 2 weeks and 3 months post treatment). For this purpose, the blood will be taken from the superficial veins of the forearm and sent for further analysis at the Medical Analytics Department of PUM in Szczecin.

ELIGIBILITY:
Inclusion Criteria:

* 1. myocardial infarction treated with primary coronary angioplasty in the last 6 months, 2. age <65 years 3. Periodontitis diagnosed according to Page criterion -

  * ≥ 2 tooth surfaces on interprimimal spaces with a loss of CAL≥4mm (not for the same tooth)
  * ≥2 tooth surface in the interpharmal space with PD≥4mm
  * positive bleeding on probing test (BOP) 4. signed informed consent

Exclusion Criteria:

1. Acute inflammation of the airways or urinary tract
2. Neoplasmas
3. Rheumatic diseases
4. Autoimmune diseases
5. Chronic liver disease
6. Chronic kidney failure 4. and 5. stage
7. History of a stroke or TIA
8. Lack of consent for participation in the study
9. Antibiotic therapy in the last 12 months
10. Periodontal treatment in the last 6 months
11. Participation in other studies

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
PD | up to 3 months
  periodontal pocket depht
Bacterial count | up to 3 months
  level in periodontal pocket
hsCRP | up to 3 months
  level in serum

SECONDARY OUTCOMES:
CAL | december 2019
  clinical attachment level
BOP | up to 3 months
  bleeding on probing
elastase | up to 3 months
  level in serum and gingival fluid
fibrynogen | up to 3 months
  level in serum
Il-6 | up to 3 months
  level in serum and gingival fluid
glucose | up to 3 months
  level in serum
HDL | up to 3 months
  level in serum
LDL | up to 3 months
  level in serum
TCH | up to 3 months
  level in serum
TG | up to 3 months
  level in serum
AST | up to 3 months
  level in serum
ALT | up to 3 months
  level in serum
GCF | up to 3 months
  gingival cervicular fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Departament of Periodontology, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No
Documentation of study participants in paper form will be kept at the Department of Periodontology. We provide information on aggregate results in tables and statistical analysis after contact by email.

REFERENCES:
- [Derived] Samulak R, Suwala M, Dembowska E. Nonsurgical periodontal therapy with/without 980 nm diode laser in patients after myocardial infarction: a randomized clinical trial. Lasers Med Sci. 2021 Jul;36(5):1003-1014. doi: 10.1007/s10103-020-03136-6. Epub 2020 Sep 4. PMID 32885341